CLINICAL TRIAL: NCT06732050
Title: Influence of Intraoperative Nociception Guided Analgesia on Perioperative Analgesia Consumption in Patients Undergoing Laparoscopic Resection of Endometriosis
Brief Title: Influence of Intraoperative Nociception Guided Analgesia on Perioperative Total Analgesic Requirement Endometriosis
Acronym: ENDONOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Urs Zingg (Other)
Responsible Party: Sponsor-Investigator, Prof Urs Zingg, Prof. Dr. med. Urs Zingg, Spital Limmattal Schlieren
Organization: Spital Limmattal Schlieren (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024-00822
Record Dates: First submitted 2024-08-21; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Perioperative Analgesia in Endometriosis
Keywords: endometriosis surgery; perioperative analgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The control group will undergo standard treatment for laparoscopic endometriosis/adenomyosis surgery at Spital Limmattal. Although the control group will not be using NOL®-monitoring to guide analgesic requirement, the monitor will be installed with a blinded screen to investigate whether our multimodal anesthesia model is in coherence with values between 10 and 25. The anesthesia care team will not be able to see the values during surgery in order to tailor analgesic requirement only by conventional clinical judgement.
- nociception guided treatment (Experimental): For the nociception level-guided group the same standard narcosis will be applied whilst ensuring that the NOL® level value will be maintained between 10 and 25.
  Interventions: Device: nociception guided treatment

INTERVENTIONS:
Device: nociception guided treatment — For the nociception level-guided group the same standard narcosis will be applied whilst ensuring that the NOL® level value will be maintained between 10 and 25.
  Arms: nociception guided treatment

SUMMARY:
Adequate analgesia in the perioperative setting is one of the most important pillars of anesthesiology. It is generally understood that poorly managed acute postoperative pain correlates with increased morbidity, prolonged recovery periods, extended opioid utilization, and serves as a predictor for chronic pain onset . On the other hand, the overuse of opioid-based analgesics during surgery may evoke respiratory depression, constipation, nausea, sedation, and opioid-induced hyperalgesia . Thus far, the lack of an objective intraoperative pain monitor has constrained anesthesia practitioners to rely on the interpretation of physiological cues such as tachycardia, hypertonia, and lacrimation as surrogate markers of pain (3). Variability in the educational background and clinical experience among providers may predispose to either excessive or inadequate administration of analgesics, consequently allowing for unfavorable postoperative outcomes. However, recent advancements have introduced novel devices for nociception measurement. Thus, a quantifiable assessment of nociception has become feasible. The most widely approved device is the Nociception Level (NOL®) index developed by Medasense in Israel. This index operates by discerning various sympathetic responses of the body to nociceptive stimuli and has been thoroughly tested on opioid-based analgesic regimens. The NOL® index uses a multiparametric approach including a random forest algorithm to measure the balance between sympathetic and parasympathetic system activity. Recently, a strong correlation has been reported between the response of the NOL® index and analgesia during surgery.

Patients being scheduled for endometriosis surgery do have a significant history of chronic pain thus being more prone to postoperative complications and therefore will benefit the most from a tailored analgesic regimen.

DETAILED DESCRIPTION:
Adequate analgesia in the perioperative setting is one of the most important pillars of anaesthesiology. It is generally understood that poorly managed acute postoperative pain correlates with increased morbidity, prolonged recovery periods, extended opioid utilization, and serves as a predictor for chronic pain onset. On the other hand, the overuse of opioid-based analgesics during surgery may evoke respiratory depression, constipation, nausea, sedation, and opioid-induced hyperalgesia. Thus far, the lack of an objective intraoperative pain monitor has constrained anaesthesia practitioners to rely on the interpretation of physiological cues such as tachycardia, hypertonia, and lacrimation as surrogate markers of pain. Variability in the educational background and clinical experience among providers may predispose to either excessive or inadequate administration of analgesics, consequently allowing for unfavorable postoperative outcomes. However, recent advancements have introduced novel devices for nociception measurement. Thus, a quantifiable assessment of nociception has become feasible. The most widely approved device is the Nociception Level (NOL®) index developed by Medasense in Israel. This index operates by discerning various sympathetic responses of the body to nociceptive stimuli and has been thoroughly tested on opioid-based analgesic regimens. The NOL® index uses a multiparametric approach including a random forest algorithm to measure the balance between sympathetic and parasympathetic system activity. Recently, a strong correlation has been reported between the response of the NOL® index and analgesia during surgery.

Patients being scheduled for endometriosis surgery do have a significant history of chronic pain thus being more prone to postoperative complications and therefore will benefit the most from a tailored analgesic regimen. Patients' existing analgesic regimen, typically comprising Paracetamol, NSAIDs, and Metamizol, will be carefully documented during preoperative anesthetic consultations and taken into account in the study protocols.

Preoperatively, patients will be staged by their gynecologists using the ENZIAN classification. The ENZIAN classification is a diagnostic system for endometriosis that covers various localizations and forms of the disease. It enables a standardized assessment for both non-invasive and invasive diagnostic procedures. The classification considers specific compartments and uses standardized coding for the severity and location of lesions. The classification is performed preoperatively using ultrasound diagnostics as well as intraoperatively and is annotated with the lower-case letters: (s)= Surgical, (u)= Ultrasound (Keckstein J, 2021). Thereby, a comprehensive picture of the disease is obtained. Deeply infiltrating endometriosis requires a more invasive procedure, a longer operating time and a higher consumption of analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Premenopausal females
* Undergoes any type of laparoscopic surgery for suspected endometriosis or adenomyosis (diagnostic/therapeutic and/or hysterectomy)

Exclusion Criteria:

* Age < 18 years
* Patients with contraindications for opioids and/or ketamine/clonidine (standard medications)
* Pregnant or breastfeeding women
* Lack of ability to follow the study procedure, e.g. due to severe language barriers, mental disorders, dementia
* Patients requiring preoperative or postoperative treatment in the intensive care unit
* Patients with conditions precluding the use of the NOL® sensor, such as neuromuscular deficits affecting hand function
* Regular consumption of opioids (Mankoski Score ≥6)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Total analgestic requirement | Start of anaesthesia until discharge from the recovery room (max. lenghth of stay in the recovery 2 hours)..
  Total analgesic requirement. Intra- and postoperative medication administration will be systematically documented throughout until two hours after arrival at the recovery room or until the patient has been discharged from the recovery room.

SECONDARY OUTCOMES:
Postoperative Numeric Rating Scale (NRS) scores in PACU | Start Start at arrival in the recovery room until discharge from the recovery room (max. lenghth of stay in the recovery 2 hours)
  Postoperative Numeric Rating Scale (NRS) scores. The NRS icludes values from 0 to 10 (indicating no pain at 0 and maximized pain at 10, which is a worse outcome). The NRS score will be assessed every 15 minutes starting with arrival at the recovery room until 2 hours after admission or until the patient has been discharged from the recovery room.
Total length of Stay in the PACU (min) | Start at arrival in the recovery room until discharge from the recovery room (max. lenghth of stay in the recovery 2 hours)
Postoperative Numeric Rating Scale (NRS) scores at discharge | Immediately postoperatively until discharge (1-3 days).
  Postoperative Numeric Rating Scale (NRS) scores at discharge (indicating no pain at 0 and maximized pain at 10, which is a worse outcome) will be assessed every 15 minutes starting with arrival at the recovery room until 2 hours after admission or until the patient has been discharged from the recovery room. One more NRS assessement will be made at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Marcolino, Dr. med., Principal Investigator — Spital STS AG
Locations (1):
- Spital Limmattal, Schlieren, Canton of Zurich, Switzerland